CLINICAL TRIAL: NCT02523716
Title: Effect of Short-term Simulated Altitude Exposure on Cardiopulmonary Functional Capacity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to maintain access to Altitude Facility
Sponsor: University of Limerick (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2014_02_33
Record Dates: First submitted 2015-06-02; First posted 2015-08-14 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2021-04

CONDITIONS: Hypoxia
Keywords: Hypoxic conditioning; Cardio pulmonary exercise testing
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypoxia (Experimental): Mild hypoxia of 15% oxygen, equivalent altitude of 2440m over a period of 7 days
  Interventions: Other: Hypoxia
- Normoxia (Sham Comparator): Exposure to normal, sea-level air
  Interventions: Other: Normoxia

INTERVENTIONS:
Other: Hypoxia — Participants live within an altitude residence facility. Hypoxic acclimatisation will be achieved by venting the rooms with air containing a reduced oxygen content. The degree of hypoxia is ramped over a 2-day period as participants experience 14 hours of overnight hypoxic exposure (simulating altitude of : 1830m on Day 1; 2130m on Day 2). The final 5 days will be spent entirely in the altitude residence facility at a consistent hypoxia level (simulating approximately 2440m).
  Arms: Hypoxia
Other: Normoxia — Participants will live in the altitude residence facility. As a sham-control, normal sea level air will be circulated throughout the house.
  Arms: Normoxia

SUMMARY:
To determine if exposure of older volunteers, age 50-70y, who are healthy, but not physically active, to 7 days of mild hypoxia (15% oxygen, equivalent 2440m) will improve cardiopulmonary functional capacity.

DETAILED DESCRIPTION:
Background There is an urgent need to reduce morbidity and mortality following major surgery. Bodily demands for oxygen increase after major surgery, and postoperative outcomes can be predicted by quantifying the body's ability to meet increased mitochondrial demand for oxygen using cardiopulmonary exercise testing (CPET).

Design This is a preliminary, physiological study to establish the baseline relationship between mild hypoxia exposure and cardiopulmonary function. This study will begin to examine the feasibility and potential for achieving risk modification through low-oxygen (hypoxic) conditioning, in which a safe and convenient "dose" of mild hypoxia is used to improve CPET derived variables that predict mortality following surgery.

The study will use a randomised, double blind, sham-controlled, crossover design. After a baseline CPET test, participants will be exposed to 7 days of either mildly hypoxic or normoxic air. A follow up CPET test will then be used to determine if cardiopulmonary functional capacity increased after exposure. After a two week washout period, participants will return for a second 7-day session where the alternate exposure will be given. A final follow-up CPET test will then be performed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female individuals aged 50-70 years with sedentary lifestyles.

Exclusion Criteria:

* Known intolerance to altitude identified by the participant's clinical examination, history and pre-altitude screening completed by the research clinician.
* Non-availability and/or suitability to complete the required residential period within the altitude centre.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Cardio pulmonary functional variables | Change in Cardio pulmonary functional variables between day 0 and day 7 in each arm of the study.
  Assess cardio pulmonary functional variables using cardio pulmonary exercise testing (CPET) prior and following participants completing each arm of the study

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Smith (Chief Investigator), MBBS, DPhil, FRCA, FAsMA, Principal Investigator — University of Oxford; Phillip Jakeman, BSc, MSc, PhD, Principal Investigator — University of Limerick